CLINICAL TRIAL: NCT00102882
Title: Randomized, Double-Blind Comparison of Advair 100/50 BID vs Salmeterol BID vs Albuterol QID in Subjects With ARG/ARG Genotype 12 Years of Age and Older With Presistent Asthma on Short-Acting Beta2-Agonists Alone
Brief Title: Study Of Asthma And Genetics In Patients To Be Treated With Fluticasone Propionate/Salmeterol Or Salmeterol Xinafoate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SFA100062
Record Dates: First submitted 2005-02-03; First posted 2005-02-04 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Asthma
Keywords: genotype; Salmeterol; ADVAIR
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination; Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: fluticasone propionate/salmeterol
Drug: salmeterol xinafoate
  Other Names: fluticasone propionate/salmeterol

SUMMARY:
This study may last up to 36-38 weeks. Patients will visit the clinic 11 times. A blood sample will be taken at Visit 1 to look at subjects' genes. Breathing tests will be done during the study. Study medicines and procedures will be provided at no cost. Patients will be treated with VENTOLIN (8 wks), ATROVENT (8 wks), then ADVAIR or SEREVENT (16 wks). ADVAIR and SEREVENT are FDA approved for the treatment of asthma in patients 4 years of age and older.

DETAILED DESCRIPTION:
A Randomized, Parallel Group, Double-Blind, Comparative Trial Assessing Lung Function and Other Measures of Asthma Control in Adults and Adolescents, at least 12 Years of Age, with Persistent Asthma, Who Have Either a B16-Arg/Arg, a B16-Gly/Gly or a B-16 Arg/Gly Genotype and are Treated With Fluticasone Propionate/Salmeterol DISKUS™ Combination Product 100/50mcg or Salmeterol DISKUS 50 mcg BID

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of persistent asthma for 3 months.
* Use of short-acting beta-agonist medication like VENTOLIN.

Exclusion criteria:

* Hospitalization for asthma 6 months before study.
* Other serious diseases like congestive heart failure, uncontrolled hypertension, TB.
* Current use of inhaled or oral corticosteroids.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2004-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Evaluate lung function by testing morning peak expiratory flow in patients with a B16 Arg/Arg genotype compared to patients with a B16 Gly/Gly genotype over 16 weeks of treatment with ADVAIR or SEREVENT

SECONDARY OUTCOMES:
Evaluate lung function by testing morning peak expiratory flow in patients with a Arg/Gly genotype compared to patients with a Arg/Arg or a Gly/Gly genotype over 16 weeks of treatment with ADVAIR and/or SEREVENT

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (78):
- United States (73):
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Inglewood, California
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Stockton, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Lakewood, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Waterbury, Connecticut
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, South Miami, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Lilburn, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Warrensburg, Missouri
  - GSK Investigational Site, Papillion, Nebraska
  - GSK Investigational Site, Hackensack, New Jersey
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Bay Shore, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Upland, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Corsicana, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Kerrville, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Bellingham, Washington
  - GSK Investigational Site, Kirkland, Washington
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
  - GSK Investigational Site, West Allis, Wisconsin
- GSK Investigational Site, Nairobi, Kenya
- Peru (2):
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, San Isidro, Lima region
- Puerto Rico (2):
  - GSK Investigational Site, Hato Rey, Puerto Rico
  - GSK Investigational Site, Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Bleecker ER, Nelson HS, Kraft M, Corren J, Meyers DA, Yancey SW, Anderson WH, Emmett AH, Ortega HG. Beta2-receptor polymorphisms in patients receiving salmeterol with or without fluticasone propionate. Am J Respir Crit Care Med. 2010 Apr 1;181(7):676-87. doi: 10.1164/200809-1511OC. Epub 2009 Nov 12. PMID 19910613
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: SFA100062 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SFA100062 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SFA100062 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SFA100062 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SFA100062 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SFA100062 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SFA100062 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register